CLINICAL TRIAL: NCT05497050
Title: The Effect of Nursing Empowerment Program Applied to Families of PKU Children, Coping Attitudes of Families and Phenylalanine Levels of Children
Brief Title: The Effect of Nursing Empowerment Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Fahri AŞKAN, PhD Candidate, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: FAHRİ AŞKAN PHD THESIS
Record Dates: First submitted 2022-08-08; First posted 2022-08-11 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Phenylketonurias
Keywords: family; Coping; Education; Phenylketonuria(PKU); Empowerment; Nursing.
MeSH Terms: conditions — Phenylketonurias; Empowerment | interventions — Sex Education

STUDY DESIGN:
Intervention Model Description: The study was completed with the families of 36 children with PKU, 19 in the intervention group and 17 in the control group, who met the inclusion criteria.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Family education
  Interventions: Behavioral: Family education
- Control group (No Intervention): No training will be given.

INTERVENTIONS:
Behavioral: Family education — By calling the families in the experimental group by phone; Nursing interventions for family empowerment will last for 10 weeks, they will be invited to the Family Health Center (FHC) or child metabolism polyclinic twice in this process, they will be called once a week (with 2 phone calls) for two weeks after the face-to-face training initiative in the first stage, In the second stage, at the end of the face-to-face training, they will be informed that they will be called once a week for two weeks (4 phone calls in total). The families in the experimental group will be informed that 4 weeks after the completion of the training and phone calls (at the 10th week), they will call the FHC or the pediatric metabolism polyclinic again for the application of the post-tests and that the nursing training for family empowerment will be completed.
  Arms: Experimental group

SUMMARY:
The study has shown that the strengthening program applied to the families of children diagnosed with phenylketonuria (PKU) and the education given; It will be conducted in order to examine the effect of the family's coping attitudes, knowledge scores about the disease and its management. The research is of the randomized controlled experimental type. Children from PKU constitute the universe in the city center of Van. The families of children between the ages of 0-3 who were diagnosed with PKU will form the sample of the study. A nursing strengthening program will be applied to families in the experimental group for 10 weeks. The scope of this program; It consists of face-to-face training on disease management, giving the educational guide (booklet) for the families of babies diagnosed with PKU, telephone calls during the education process and counseling services. No application will be made to the families in the control group. After the application of the last tests to the control group; Face-to-face training and a booklet will be given to the experimental group. Data; It will be collected with 'Child and Family Introductory Information Form', 'Parents' Information Level Assessment Form about Phenylketonuria' and 'Coping Attitudes Assessment Scale'.

In the literature, there is no study showing the effect of the education given to the families of babies diagnosed with PKU on their coping attitudes. Based on the need to fill this knowledge gap in the literature, it is thought that the study will contribute to the field of child health and disease nursing.

DETAILED DESCRIPTION:
Phenylketonuria is a disorder of phenylalanine metabolism and causes intellectual destruction if left untreated. It is an autosomal recessive metabolic disease that develops as a result of the absence of the enzyme phenylalanine hydroxylase (FAH), which provides the necessary amino acid metabolism for protein production in the body, which causes high phenylalanine in the blood. In our country, it is one of the places where PKU is commonly encountered (Çavuşoğlu, 2015; Hafid et al, 2015; Törner and Büyükgönenç, 2013). While the incidence of this disease in European countries is 1/10000-30000, it is 1/3000-4500 in our country (Alparslan, 2021). This situation is directly related to consanguineous marriages. It is stated that one out of every five marriages in our country is consanguineous marriage. If left untreated, it can cause extreme mental retardation, convulsions and death (Alparslan, 2021; Çavuşoğlu, 2015; Hafid et al, 2015; Törner and Büyükgönenç, 2013).

The care of the child with phenylketonuria is carried out by the parents. Extra care (diet therapy, control of blood phenylalanine level, etc.) for children in this diagnosis group is provided by their parents. The treatment and care process of children with PKU affects family routines, relationships and parenting styles. Parents of children experience emotional and economic burden. Therefore, it is stated that the care burden of parents in this diagnosis group is higher than that of healthy parents, and their quality of life is lower (Hatzmann et al, 2009). In addition, studies have shown that families of children with PKU have high levels of anxiety, depression (Mahmoudi-Gharaei et al. 2011) and stress (Irannejad et al. 2018). In another study; It is reported that the family's routines have changed (not eating in front of the child, not eating in restaurants, etc.) and that they experience anxiety about the effect of diet incompatibility on blood phenylalanine levels, feeling overwhelmed and guilt in the care process (Carpenter et al 2018). Therefore, having a child with PKU may affect coping attitudes.

Child health and diseases nurse should support children with PKU and their families on issues such as informing, training and counseling about the disease and its management.

ELIGIBILITY:
Inclusion Criteria:

* Residing in Van and/or being followed up in the pediatric metabolism polyclinic,
* Agreeing to participate in the research,
* literate,
* Speaking and understanding Turkish,
* 18 years old and over
* Fully oriented and cooperative and open to communication,
* a parent who is the primary caregiver of the child,
* The child is in the 0-3 age range (≤3 years old),
* Families of children with definitive diagnosis of PKU will be included.

Exclusion Criteria:

* Not residing in Van and/or not being followed up in the pediatric metabolism polyclinic,
* Those who do not accept to participate in the research, who are illiterate,
* Does not speak or understand Turkish,
* Parent/family member who is aged 17 or younger, who is not fully oriented and cooperative and not open to communication, and does not provide primary care for the child,
* The child is over 3 years old (3 years <),
* Dropping out of the training to be applied,
* Families of children with PKU who are not definitively diagnosed will not be included in the study.

Ages: 1 Day to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2021-11-24 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-06-22 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Evaluation Of Coping Attitudes (COPE) at week 10 | 10 week
  *COPE is a validated. The scale is a 4-point Likert type scale. While scoring the items, 1 point is given for "I Never Do This", 2 points for "I rarely do this", 3 points for "I do this way", and 4 points for "I Do This Mostly". There is no negative item in the scale. The highest score that can be obtained from the scale is 128, and the lowest score is 32. A high score from the scale means a high level of coping attitude, and a low score means a low level of coping attitude.
  change = (Week 10 Score - Baseline Score)

SECONDARY OUTCOMES:
Change from Baseline in Evaluation of the level of knowledge about PKU at week 1 | 10 week
  Form for Evaluation of Families' Knowledge Levels on Phenylketonuria:
  *Question form prepared by the researcher in line with the literature; The level of knowledge of families about the disease and disease management of their child with PKU will be measured. The form consists of 20 questions.The increase in the mean of correct answers obtained in the form indicates that the level of knowledge about the disease is good.
  change = (Week 10 Score - Baseline Score)

CONTACTS AND LOCATIONS:
Overall Officials: Şenay ÇETİNKAYA, Doç. Dr., Study Director — Cukurova University
Locations (1):
- Van Yuzuncu Yıl University, Van, Tuşba, Turkey (Türkiye)

REFERENCES:
- [Background] MacDonald A, Depondt E, Evans S, Daly A, Hendriksz C, Chakrapani A A, Saudubray JM. Breast feeding in IMD. J Inherit Metab Dis. 2006 Apr-Jun;29(2-3):299-303. doi: 10.1007/s10545-006-0332-x. PMID 16763891
- [Background] Pinto A, Adams S, Ahring K, Allen H, Almeida MF, Garcia-Arenas D, Arslan N, Assoun M, Atik Altinok Y, Barrio-Carreras D, Belanger Quintana A, Bernabei SM, Bontemps C, Boyle F, Bruni G, Bueno-Delgado M, Caine G, Carvalho R, Chrobot A, Chyz K, Cochrane B, Correia C, Corthouts K, Daly A, De Leo S, Desloovere A, De Meyer A, De Theux A, Didycz B, Dijsselhof ME, Dokoupil K, Drabik J, Dunlop C, Eberle-Pelloth W, Eftring K, Ekengren J, Errekalde I, Evans S, Foucart A, Fokkema L, Francois L, French M, Forssell E, Gingell C, Goncalves C, Gokmen Ozel H, Grimsley A, Gugelmo G, Gyure E, Heller C, Hensler R, Jardim I, Joost C, Jorg-Streller M, Jouault C, Jung A, Kanthe M, Koc N, Kok IL, Kozanoglu T, Kumru B, Lang F, Lang K, Liegeois I, Liguori A, Lilje R, Lubina O, Manta-Vogli P, Mayr D, Meneses C, Newby C, Meyer U, Mexia S, Nicol C, Och U, Olivas SM, Pedron-Giner C, Pereira R, Plutowska-Hoffmann K, Purves J, Re Dionigi A, Reinson K, Robert M, Robertson L, Rocha JC, Rohde C, Rosenbaum-Fabian S, Rossi A, Ruiz M, Saligova J, Gutierrez-Sanchez A, Schlune A, Schulpis K, Serrano-Nieto J, Skarpalezou A, Skeath R, Slabbert A, Straczek K, Gizewska M, Terry A, Thom R, Tooke A, Tuokkola J, van Dam E, van den Hurk TAM, van der Ploeg EMC, Vande Kerckhove K, Van Driessche M, van Wegberg AMJ, van Wyk K, Vasconcelos C, Velez Garcia V, Wildgoose J, Winkler T, Zolkowska J, Zuvadelli J, MacDonald A. Weaning practices in phenylketonuria vary between health professionals in Europe. Mol Genet Metab Rep. 2018 Nov 25;18:39-44. doi: 10.1016/j.ymgmr.2018.11.003. eCollection 2019 Mar. PMID 30705824
- [Background] van Spronsen FJ, Blau N, Harding C, Burlina A, Longo N, Bosch AM. Phenylketonuria. Nat Rev Dis Primers. 2021 May 20;7(1):36. doi: 10.1038/s41572-021-00267-0. PMID 34017006